CLINICAL TRIAL: NCT04681859
Title: Safety and Efficacy Evaluation of a Low-cost CPAP Device for Hypoxemic COVID-19 Patients: A Pilot Study
Brief Title: Evaluation of a Low-cost CPAP Device on Hospitalized COVID-19 Patients
Acronym: OxyJet-CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh University of Engineering and Technology (Other)
Collaborators: Dhaka Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BME-BUET-003
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Hypoxemia
MeSH Terms: conditions — COVID-19; Hypoxia | interventions — Therapeutics; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Oxygen (HFNO) treatment (Active Comparator)
  Interventions: Device: High Flow Nasal Oxygen (HFNO) treatment
- Continuous positive airway pressure (CPAP) therapy using OxyJet (Experimental)
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) therapy using OxyJet

INTERVENTIONS:
Device: High Flow Nasal Oxygen (HFNO) treatment — Administration of High Flow Nasal Oxygen (HFNO) to patients who did not respond to standard low-flow oxygen therapy (non-rebreather mask on 15L/min). Adjust flow-rate and FiO2 as per standard HFNO treatment protocol.
  Arms: High Flow Nasal Oxygen (HFNO) treatment
Device: Continuous Positive Airway Pressure (CPAP) therapy using OxyJet — Administer CPAP to patients who did not respond to standard low-flow oxygen therapy (non-rebreather mask on 15L/min). CPAP initiated with FiO2 at 40% and a 10cm PEEP. Titrate PEEP to 15 cm if required. Deliver additional oxygen via secondary port if a higher FiO2 is required.
  Arms: Continuous positive airway pressure (CPAP) therapy using OxyJet

SUMMARY:
The aim of this study is to evaluate the preliminary safety and performance of a low-cost locally-made Venturi-based Non-invasive Positive Pressure Ventilator (NIPPV) device for hypoxemic COVID-19 patients. The device administers Continuous Positive Airway Pressure (CPAP) therapy using the jet-mixing or Venturi effect to increase the volume flow rate of oxygenated air from a pressurized cylinder by entraining the atmospheric air. To provide CPAP therapy, this high flow of oxygenated air is delivered to the patient via a low-cost non-vented mask with a tight seal with a High-Efficiency Particulate Air (HEPA) filter connected to the exhalation limb. The tight seal and HEPA filter ensures a minimal risk of aerosol generation and thus the device can be used without a negative pressure room. The system consists of the developed Venturi-based flow-generator, a standard 22mm breathing tube, a standard Y-connector, a non-vented CPAP mask (e.g., snorkel mask, helmet), a HEPA filter, and a Positive End Expiratory Pressure (PEEP) valve. The bench-top testing of the device is done in the laboratories of BUET and was verified that the device performs within the CPAP guidelines provided by the Medicines and Healthcare products Regulatory Agency (MHRA), UK. This study aims to assess the safety of and efficacy of the device in three different steps: (1) design validation, (2) clinical feasibility and (3) pilot clinical trial for safety and efficacy evaluation. Only if the device successfully passes the parts 1 and 2, the investigators will proceed to the final clinical trial in step 3. In this final step, the investigators aim to conduct a randomized controlled trial (RCT) evaluating for non-inferiority of the CPAP intervention compared to standard HFNO treatment. The number of ventilator-free days will be used as the primary outcome for efficacy, while patient recovery, death, or need of intubation and other adverse events will be used as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed or suspected COVID-19 patient (by RT-PCR) having severe pneumonia and hypoxemia (SpO2 ≤90%) who did not respond to standard oxygen therapy (non-rebreather mask on 15L/min at 100% FiO2).

Exclusion Criteria:

* Severely hypoxemic patients (SpO2≤85%)
* Patients with low respiratory drive or requiring cardiopulmonary resuscitation
* Patients with contraindications for CPAP
* Pregnant status
* Age > 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days | 10 days
  The total number of days the patient was able to avoid being placed under a mechanical ventilator.

SECONDARY OUTCOMES:
Recovery of the patient | 30 days
  The event that the patient has recovered and released from the hospital within 30 days.
Death or need of intubation | 10 days
  The event that the patient dies or requires to be placed under a mechanical ventilator.
Oxygen toxicity or other adverse events | 10 days
  Oxygen toxicity or other adverse event rating according to the CTCAE scale (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Taufiq Hasan, PhD, Principal Investigator — Bangladesh University of Engineering and Technology; Dr. Robed Amin, MBBS, FCPS, Principal Investigator — Dhaka Medical College
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No